CLINICAL TRIAL: NCT06841133
Title: The Effectiveness of Chinese Art Activities Combined With Peer Group Participation on Psychological Well Being Among Newly Old Chinese of Elderly Center: Randomized Controlled Trail
Brief Title: Chinese Art Activities or Combined With Peer Group Participation on Psychological Well Being
Acronym: CAA+PGP#PWB
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Prince of Songkla University (Other)
Responsible Party: Principal Investigator, Liping Pu, Principal Investigator, Prince of Songkla University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: PSU IRB 2024-St-Nur 048
Record Dates: First submitted 2025-02-08; First posted 2025-02-24 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-02

CONDITIONS: Aging
Keywords: Art Activity; Peer Group; psychological well-being; older
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Chinese Art Activities (CAA) (Experimental): Participants will receive routine care plus the CAA intervention. The intervention is delivered over three sessions within one week (day1,3,5), with each session lasting 50 minutes.Baseline measures are collected pre-randomization. Outcomes are assessed 30 minutes before and after each intervention session . A final follow-up assessment is conducted one week after the last intervention.
  Interventions: Behavioral: Chinese Art Activities
- Chinese Art Activities combined with Peer Group Participation (PGP) (Experimental): Participants will receive routine care plus the CAA and PGP intervention. The intervention is delivered over three sessions within one week (day1,3,5), with each session lasting 80 minutes.Baseline measures are collected pre-randomization. Outcomes are assessed 30 minutes before and after each intervention session . A final follow-up assessment is conducted one week after the last intervention
  Interventions: Behavioral: Chinese Art Activities combined with Peer Group Participation (PGP)
- routine care (No Intervention): Participants in both the intervention and control groups will receive identical routine care, including daily activities such as simple limb exercises and group walks.

INTERVENTIONS:
Behavioral: Chinese Art Activities — This activity based on Recreation therapy, aims to heal the psychological symptom cluster and enhance the PWB of the old Chinese transit to the elderly center. The activity follows the usual care during the process with the addition of Chinese art activities. It employed the following two main activities:
  (1) Traditional Chinese landscape painting; (2) Calligraphy. The activity will be conducted 50min by researchers. It can be conducted at hall, conference room, etc. in the elderly center (EC), and it is a group intervention
  Arms: Chinese Art Activities (CAA)
Behavioral: Chinese Art Activities combined with Peer Group Participation (PGP) — The activity follows the usual care during the process with the addition of Chinese art activities combined with Peer Group Participation. The activity will be conducted 80min by researchers. In groups of 5 people, after the painting and calligraphy activity, under the organization of peers, each group member will show their works and talk about their feelings and views on their works. They will also share the reasons why they chose these words or sentences. Everyone must say words of comfort and encouragement to others' work.
  Arms: Chinese Art Activities combined with Peer Group Participation (PGP)

SUMMARY:
The goal of this trial is to evaluate the effects of two interventions : routine care plus Chinese Art Activities(+CAA) and routine care plus Chinese Art Activities combined with Peer Group Participation (+CAA+PGP) on psychological well-being, loneliness, happiness, relaxation, and salivary cortisol levels in elderly participants (aged 60-85, new residents with ≤1 year of stay). The main questions it aims to answer are:

* Does the +CAA intervention improve psychological well-being and related outcomes compared to routine care?
* Does the +CAA+PGP intervention provide additional benefits over +CAA alone? Researchers will compare three groups (Group A: +CAA, Group B: +CAA +PGP, Group C: routine care) to see if the interventions lead to immediate and sustained improvements in the measured outcomes.

Participants will:

* Undergo baseline assessments of psychological well-being(PWB), loneliness, happiness, relaxation, and salivary cortisol levels.
* Receive their assigned intervention over three sessions within one week (Monday, Wednesday, Friday).
* Complete outcome measures 30 minutes before and after each session.
* Participate in a final follow-up assessment one week after the last session to evaluate sustained effects.

DETAILED DESCRIPTION:
This multi-center, randomized, assessor-blind trial is designed based on the Max.-Min.-Con. principle, which aims to maximize the benefits of the intervention while minimizing potential confounding factors and ensuring control over the study design. The trial features three parallel intervention groups: control (routine care), +CAA, and +CAA+PGP, with a 1:1:1 allocation ratio. This balanced allocation ensures that each intervention group and the control group have an equal number of participants, allowing for a fair comparison of outcomes.

The study is conducted sequentially across three elderly centers, with each center serving as an independent randomization unit. This multi-center approach enhances the generalizability of the findings by including diverse populations from different locations. Within each institution, 30 participants (aged 60-85, new residents with ≤1 year of stay) are recruited through health providers, totaling 90 elderly participants across all three centers. The inclusion of new residents (with ≤1 year of stay) is critical, as this population is particularly vulnerable to stress and reduced psychological well-being (PWB) during the transition to elderly care centers.

To ensure balanced groups and control for confounding variables, minimized randomization is employed. Within each institution, the 30 participants are divided into three groups-Group A, Group B, and Group C-with 10 participants in each group. Group A receives the +CAA intervention, Group B receives the +CAA+PGP intervention, and Group C serves as the control group, receiving only routine care. The use of minimized randomization helps to balance key confounding factors such as age and visitation frequency, ensuring that the groups are comparable at baseline.

The intervention is delivered over three sessions within one week, specifically on day 1, day 3 and day 5. This schedule allows for consistent exposure to the interventions while providing adequate time for participants to rest between sessions. The +CAA intervention involves traditional Chinese art activities, such as calligraphy and painting, which are designed to promote relaxation and emotional well-being. The +CAA+PGP intervention** builds on this by incorporating peer group discussions, where participants share their experiences and artworks, fostering social interaction and mutual support.

Baseline assessments of key outcomes-psychological well-being (PWB), loneliness, happiness, relaxation, and salivary cortisol levels-are conducted prior to randomization. These baseline measures provide a reference point for evaluating the impact of the interventions. To capture the immediate effects of the interventions, outcome measures are collected 30 minutes before and after each intervention session. This allows the researchers to assess short-term changes in PWB, emotional states, and stress levels (as indicated by salivary cortisol).

Additionally, a final follow-up assessment is conducted one week after the last intervention session to evaluate the sustained outcomes of the interventions. This follow-up assessment is crucial for determining whether the benefits of the interventions persist beyond the immediate post-intervention period.

In summary, this trial is designed to rigorously evaluate the effectiveness of Chinese Art Activities (CAA) and their combination with Peer Group Participation (PGP) in improving psychological well-being and reducing stress among elderly residents transitioning to care centers. By employing a multicenter, randomized, and assessor-blind design, the study ensures robust and reliable results that can inform future interventions in elderly care settings.

ELIGIBILITY:
Inclusion Criteria:

* Age 60-85 years.
* Older persons living in Elderly Centers (ECs) for the first time, with a duration of stay ≤1 year.
* Normal cognitive function (Mini-Mental State Examination [MMSE] score >24).
* Possess necessary reading and writing skills.
* Volunteer to participate in the study.

Exclusion Criteria:

* Older persons with serious diseases (e.g., heart failure, asthma, cerebrovascular disease, advanced tumors).
* Older persons who later leave the elderly center.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-07-09 (Estimated); Primary Completion 2025-07-19 (Estimated); Study Completion 2025-08-09 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Psychological Well-Being (PWB) Score at End of Intervention | From enrollment to one week after the final intervention session
  Psychological well-being was assessed using the 18-item Chinese version of Ryff's Psychological Well-Being Scale. This scale measures six dimensions of well-being: autonomy, environmental mastery, personal growth, positive relations with others, purpose in life, and self-acceptance. Each item is scored on a 6-point Likert scale (1=strongly disagree, 6=strongly agree). The total score ranges from 18 to 108, with higher scores indicating better psychological well-being.
Change From Baseline in Happiness Score at End of Intervention | From enrollment to one week after the final intervention session
  Happiness was measured using a 100 mm Visual Analog Scale (VAS). Participants were asked to mark their current level of happiness on a horizontal line, where 0 mm represents "not happy at all" and 100 mm represents "extremely happy." The VAS is a widely used tool for assessing subjective feelings, and higher scores indicate greater happiness.
Change From Baseline in Relaxation Score at End of Intervention | From enrollment to one week after the final intervention session
  Relaxation was measured using a 100 mm Visual Analog Scale (VAS). Participants were asked to mark their current level of relaxation on a horizontal line, where 0 mm represents "not relaxed at all" and 100 mm represents "extremely relaxed." The VAS is a validated tool for assessing subjective states, and higher scores indicate greater relaxation.
Change From Baseline in Loneliness Score at End of Intervention | From enrollment to one week after the final intervention session
  Loneliness was measured using a 100 mm Visual Analog Scale (VAS). Participants were asked to mark their current level of loneliness on a horizontal line, where 0 mm represents "extremely lonely" and 100 mm represents "not lonely at all." The VAS is a reliable tool for assessing subjective feelings, and higher scores indicate lower loneliness.
Change From Baseline in Salivary Cortisol Level at End of Intervention | From enrollment to one week after the final intervention session
  Salivary cortisol levels were measured as an indicator of stress response. Participants provided saliva samples, which were analyzed in a specialized laboratory using enzyme-linked immunosorbent assay (ELISA) techniques. Cortisol levels are reported in nmol/L, and higher values may indicate higher stress levels. This method is non-invasive and widely used in stress-related research.

CONTACTS AND LOCATIONS:
Overall Officials: Liping Pu, Principal Investigator — Phd candidate of Faculty of Nursing Prince of Songkla University
Locations (3):
- China (3):
  - Sukangyang · Gaoxin Yiyang, Suzhou, Jiangsu
  - Sukangyang · Jiangling, Suzhou, Jiangsu
  - Sukangyang · Yiyang, Suzhou, Jiangsu

IPD SHARING:
Plan to Share IPD: Yes
The corresponding author's contact details will be publicly available for researchers to contact the investigators. Data are available upon written request, in accordance with the General Data Protection Regulation (GDPR)
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After finishing the research
Access Criteria: Data are available upon written request, in accordance with the General Data Protection Regulation (GDPR)

REFERENCES:
- [Background] Aydin M, Kutlu FY. The Effect of Group Art Therapy on Loneliness and Hopelessness Levels of Older Adults Living Alone: A Randomized Controlled Study. Florence Nightingale J Nurs. 2021 Oct;29(3):271-284. doi: 10.5152/FNJN.2021.20224. PMID 35110167
- [Background] Bourdon E, Belmin J. Enriched gardens improve cognition and independence of nursing home residents with dementia: a pilot controlled trial. Alzheimers Res Ther. 2021 Jun 16;13(1):116. doi: 10.1186/s13195-021-00849-w. PMID 34134758
- [Background] Ellis JM. Psychological transition into a residential care facility: older people's experiences. J Adv Nurs. 2010 May;66(5):1159-68. doi: 10.1111/j.1365-2648.2010.05280.x. PMID 20423358
- [Background] Hermann C. Bonsai as a group art therapy intervention among traumatized youth in KwaZulu-Natal. Psych J. 2021 Apr;10(2):177-186. doi: 10.1002/pchj.440. Epub 2021 Mar 9. PMID 33751848
- [Background] Koppitz AL, Dreizler J, Altherr J, Bosshard G, Naef R, Imhof L. Relocation experiences with unplanned admission to a nursing home: a qualitative study. Int Psychogeriatr. 2017 Mar;29(3):517-527. doi: 10.1017/S1041610216001964. Epub 2016 Nov 17. PMID 27852339
- [Background] Lan X, Xiao H, Chen Y. Life review for Chinese older adults in nursing homes: cultural acceptance and its effects. Int Psychogeriatr. 2019 Apr;31(4):527-535. doi: 10.1017/S1041610218001084. Epub 2018 Oct 2. PMID 30277193
- [Background] Mello S, O'Connor KA. Morbidity and Mortality Following Relocation of Highly Dependent Long-Term Care Residents: A Retrospective Analytical Study. J Gerontol Nurs. 2016 Nov 1;42(11):34-38. doi: 10.3928/00989134-20160908-01. Epub 2016 Oct 5. PMID 27711930
- [Background] Rebok GW, Ball K, Guey LT, Jones RN, Kim HY, King JW, Marsiske M, Morris JN, Tennstedt SL, Unverzagt FW, Willis SL; ACTIVE Study Group. Ten-year effects of the advanced cognitive training for independent and vital elderly cognitive training trial on cognition and everyday functioning in older adults. J Am Geriatr Soc. 2014 Jan;62(1):16-24. doi: 10.1111/jgs.12607. Epub 2014 Jan 13. PMID 24417410
- [Background] Sun C, Yu Y, Li X, Cui Y, Ding Y, Zhu S, Li X, Chen S, Zhou R. The factors of adaptation to nursing homes in mainland China: a cross-sectional study. BMC Geriatr. 2020 Nov 30;20(1):517. doi: 10.1186/s12877-020-01916-x. PMID 33256628
- [Background] Sun C, Zhou R, Cui Y, Ding Y, Li X, Li X, Zhang Y, Chen S, Xing Y. The Adaptation of Older Adults' Transition to Nursing Homes in Mainland China: A Qualitative Study. J Transcult Nurs. 2021 Jul;32(4):318-325. doi: 10.1177/1043659620923387. Epub 2020 May 23. PMID 32449461
- [Background] Wu CS, Rong JR. Relocation experiences of the elderly to a long-term care facility in Taiwan: a qualitative study. BMC Geriatr. 2020 Aug 6;20(1):280. doi: 10.1186/s12877-020-01679-5. PMID 32762717